CLINICAL TRIAL: NCT04675034
Title: A Randomised, Double-blind, Placebo-controlled, Dose-response Study of the Efficacy and Safety of MEDI7352 in Subjects With Painful Osteoarthritis of the Knee
Brief Title: A Study of the Efficacy and Safety of MEDI7352 in Participants With Painful Osteoarthritis of the Knee
Acronym: BESPOKE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5680C00003; 2020-003797-51 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-12-19 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Painful Osteoarthritis of the Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is a Phase IIb, multinational, multicentre, randomised, double-blind, placebo-controlled, dose-response study of MEDI7352 in participants 18 to 80 years of age (inclusive) with moderate-to-severe chronic pain of the knee. The study consists of a screening period of up to 45 days, a 12-week treatment period, and a 24-week follow-up (FU) period.
  Daily pain scores (as measured on an 11-point numerical rating scale [NRS]) recorded at the first screening visit and from Day -7 to Day -1 will be used be used to determine eligibility.
  Participants will be randomised to one of 4 doses of MEDI7352 or placebo. Each participant will receive 6 doses of MEDI7352 or placebo during the treatment period.
  After the end-of-treatment (EOT) visit at Week 12, participants will enter the FU period, which comprises 3 clinic visits (Weeks 18, 32, and 36) and 4 FU phone calls (Weeks 15, 21, 24, and 28). All participants who receive investigational product (IP) are expected to complete the FU period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be centrally assigned to randomised IP using an Interactive Response Technology/Randomisation and Trial Supply Management (IRT/RTSM) system. Before the study is initiated, telephone number and call-in directions for IRT and/or log in information and directions for RTSM will be provided to each site.
  The IRT/RTSM will provide investigator(s) or appropriate study personnel with kit identification number to be allocated to participant at IP dosing visit.
  Details for this will be described in IRT/RTSM user manual that will be provided to each centre.
  All participants, investigators, and study personnel involved in conduct of the study will be blinded to treatment assignment. The unblinded study personnel (eg, site pharmacist) will not participate in study procedures or data analysis prior to unblinding of study data to all study-related personnel. Unblinded AstraZeneca personnel who are not otherwise involved in study will prepare data for review and interim analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MEDl7352 Dose 1 (Experimental): Participants received 6 doses of subcutaneous (SC) MEDl7352 Dose 1 injection once every 2 weeks (Q2W) during a 12-week parallel-group treatment period.
  Interventions: Drug: MEDI7352
- MEDl7352 Dose 2 (Experimental): Participants received 6 doses of SC MEDl7352 Dose 2 injection Q2W during a 12-week parallel-group treatment period.
  Interventions: Drug: MEDI7352
- MEDl7352 Dose 3 (Experimental): Participants received 6 doses of SC MEDl7352 Dose 3 injection Q2W during a 12-week parallel-group treatment period.
  Interventions: Drug: MEDI7352
- MEDl7352 Dose 4 (Experimental): Participants received 6 doses of SC MEDl7352 Dose 4 injection Q2W during a 12-week parallel-group treatment period.
  Interventions: Drug: MEDI7352
- Placebo (Placebo Comparator): Participants received 6 doses of SC placebo injection matched to MEDl7352 Q2W during a 12-week parallel-group treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MEDI7352 — Participants will receive SC injection of MEDI7352 as stated in arm description.
  Arms: MEDl7352 Dose 1; MEDl7352 Dose 2; MEDl7352 Dose 3; MEDl7352 Dose 4
Other: Placebo — Participants will receive SC injection of placebo as stated in arm description.
  Arms: Placebo

SUMMARY:
This is a Phase IIb randomised, double-blind, placebo-controlled, dose-response study in participants with painful osteoarthritis (OA) of the knee. The study will assess the safety and efficacy of multiple doses of MEDI7352 compared to placebo, as well as the pharmacokinetics, pharmacodynamics and immunogenicity of MEDI7352 in participants with moderate to severe chronic pain persistent for 3 months or more not adequately controlled by standard of care treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must understand the nature of the study and must give signed and dated written informed consent prior to the initiation of any study procedures, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. For participants participating in the optional genetic research, a separate signed and dated optional genetic research ICF must be provided prior to collection of samples for optional genetic research that supports the Genomics Initiative. If a participant declines to participate in the genetic research, this will have no influence on the ability of a participant to participate in the study.
3. The participant should be willing and able to understand and comply with all protocol-specified restrictions and procedures and be able to use an electronic patient-reported outcome (ePRO) device as judged by the investigator.
4. The participant must be considered likely to comply with the study protocol and to have a high probability of completing the study, as judged by the investigator.
5. The participant must be willing and able to discontinue all analgesic therapy with nonsteroidal anti-inflammatory drugs (NSAID) or cyclooxygenase-2 (COX-2) inhibitors from the start of the washout period until the end of the FU period. This includes over-the-counter (OTC) pain medications and topical analgesics that contain an NSAID or COX-2 inhibitor.

Exclusion Criteria:

1. Requires current treatment with another biologic therapeutic agent, disease-modifying antirheumatic drug (DMARD), or other immunosuppressants.
2. Previously received any form of anti-nerve growth factor (NGF); received anti-tumour necrosis factors (TNFs) including but not limited to golimumab, certolizumab, infliximab, adalimumab, etanercept, or rituximab within 12 months prior to screening, or other biological DMARDs (including but not limited to abatacept, tocilizumab, and tofacitinib), or other immunosuppressants within 6 months prior to screening (with the exception of inhaled or topical corticosteroids).
3. Currently receiving strong opioids for any indication.
4. Participation in another clinical study with an IP or device within 60 days or 5 half-lives, whichever is longer, prior to screening.
5. Plasma donation within 28 days of screening or any blood donation or blood loss > 500 mL within 2 months of screening.
6. Previous allogeneic bone marrow or stem cell transplant.
7. Received nonleukocyte-depleted whole blood transfusion within 120 days of the genetic research sample collection, if participating in the optional genetic research.
8. Involvement in the planning and/or conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- Research Site, Frederiksberg, Denmark
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (3):
  - Research Site, Bad Doberan
  - Research Site, Leipzig
  - Research Site, Munich
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Staszów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Zamość
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Sabadell
  - Research Site, Santiago de Compostela
  - Research Site, Santiago de Compostela-Coruña
  - Research Site, Valencia
- United Kingdom (13):
  - Research Site, Corby
  - Research Site, Enfield
  - Research Site, Glasgow
  - Research Site, High Wycombe
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Northwich
  - Research Site, Northwood
  - Research Site, Orpington
  - Research Site, Preston
  - Research Site, Rochdale
  - Research Site, Salford
  - Research Site, Shipley

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool.
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be In place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5680C00003&attachmentIdentifier=8e130b5d-6abf-4fdb-8ced-ef32e98cf47c&fileName=MEDI7352_Study_03_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 sites in 6 countries (the United Kingdom, Denmark, Estonia, Germany, Poland, and Spain).
Pre-assignment Details: A total of 345 participants were randomized, of which 344 participants received at least one dose of study drug.
Groups:
- MEDl7352 Dose Level 1: Participants received 6 doses of subcutaneous (SC) MEDl7352 Dose Level 1 injection once every 2 weeks (Q2W) during a 12-week parallel-group treatment period.
- MEDl7352 Dose Level 2: Participants received 6 doses of SC MEDl7352 Dose Level 2 injection Q2W during a 12-week parallel-group treatment period.
- MEDl7352 Dose Level 3: Participants received 6 doses of SC MEDl7352 Dose Level 3 injection Q2W during a 12-week parallel-group treatment period.
- MEDl7352 Dose Level 4: Participants received 6 doses of SC MEDl7352 Dose Level 4 injection Q2W during a 12-week parallel-group treatment period.
Period: Overall Study
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Started | 70 | 68 | 69 | 68 | 70
Treated | 70 | 68 | 69 | 68 | 69
Completed | 59 | 64 | 65 | 57 | 61
Not Completed | 11 | 4 | 4 | 11 | 9
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 9 | 3 | 4 | 8 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants analyzed according to the Intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo | Total
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 70 | 345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (7.90) | 63.3 (7.73) | 63.8 (6.91) | 63.3 (7.52) | 62.5 (8.03) | 63.7 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 51 | 48 | 46 | 42 | 230
  Male | 27 | 17 | 21 | 22 | 28 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 1 | 0 | 5
  Not Hispanic or Latino | 69 | 67 | 67 | 67 | 70 | 340
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 69 | 66 | 67 | 65 | 67 | 334
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average of Daily Numerical Rating Scale (NRS) Pain Score to Week 12
Description: Change from baseline in weekly average of daily NRS pain score to Week 12 is reported. The NRS is an 11-point Likert scale used to assess pain, where participants were asked to describe their average pain in the target knee by identifying a number from 0 = "no pain" to 10 = "most severe pain imaginable over the previous 24 hours". This was recorded on a daily basis at approximately the same time every morning via electronic patient recorded outcome (ePRO) diary. A two-step multiple imputation procedure was used to address missing post-baseline scores.
Time Frame: Baseline (Day -7 to Day -1, inclusive) through Week 12
Population: Full analysis set (FAS) included all randomized participants analyzed according to the intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 70
Unit on a scale | -2.19 (2.243) | -3.00 (2.342) | -2.83 (2.522) | -2.81 (2.835) | -2.35 (2.364)
Statistical Analysis 1: Comparison: MEDl7352 Dose Level 1 vs Placebo; Test type: Superiority; p = 0.360, ANCOVA; Least Square (LS) mean and treatment group difference with associated 95% confidence intervals (CIs) are modelled using ANCOVA on imputed data; Combined estimate for LS mean = -0.15, 95% CI 2-sided [-0.968 to 0.670], Standard Error of Mean 0.416
Statistical Analysis 2: Comparison: MEDl7352 Dose Level 2 vs Placebo; Test type: Superiority; p = 0.029, ANCOVA; Least Square mean and treatment group difference with associated 95% CIs are modelled using ANCOVA on imputed data; Combined estimate for LS mean = -0.80, 95% CI 2-sided [-1.619 to 0.027], Standard Error of Mean 0.418
Statistical Analysis 3: Comparison: MEDl7352 Dose Level 3 vs Placebo; Test type: Superiority; p = 0.026, ANCOVA; Least Square mean and treatment group difference with associated 95% CIs are modelled using ANCOVA on imputed data; Combined estimate for LS mean = -0.80, 95% CI 2-sided [-1.618 to 0.009], Standard Error of Mean 0.413
Statistical Analysis 4: Comparison: MEDl7352 Dose Level 4 vs Placebo; Test type: Superiority; p = 0.083, ANCOVA; Least Square mean and treatment group difference with associated 95% CIs are modelled using ANCOVA on imputed data; Combined estimate for LS mean = -0.59, 95% CI 2-sided [-1.423 to 0.245], Standard Error of Mean 0.424

2. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Subscale to Week 12
Description: The WOMAC multiscale index is used to assess pain, stiffness, and joint functionality in the past 48 hours in participants with OA of the knee or hip. The WOMAC pain subscale consists of 5 questions assessing the participant's pain due to osteoarthritis (OA) in the target knee. Each question was scored on a NRS scale from 0 to 10, and the WOMAC pain subscale score is calculated as the mean score from all 5 questions, where higher scores represent higher pain. Change from baseline in WOMAC pain subscale to Week 12 is reported. A two-step multiple imputation procedure was used to address missing post-baseline scores.
Time Frame: Week 0 (Day 1; baseline) through Week 12
Population: FAS included all randomized participants analyzed according to the intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 70
Unit on a scale | -1.88 (2.047) | -2.88 (2.407) | -2.62 (2.305) | -2.57 (2.992) | -2.62 (2.558)

3. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale to Week 12
Description: The WOMAC multiscale index is used to assess pain, stiffness, and joint functionality in the past 48 hours in participants with OA of the knee or hip. The WOMAC physical function (PF) subscale consists of 17 questions assessing the participant's difficulty in performing activities of daily living due to OA in the target knee. Each question is scored on an NRS scale from 0 to 10, and the WOMAC PF subscale score is calculated as the mean score from all 17 questions, where higher scores represent worse function. Change from baseline in WOMAC physical function to Week 12 is reported. A two-step multiple imputation procedure was used to address missing post-baseline scores.
Time Frame: Week 0 (Day 1; baseline) through Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 70
Unit on a scale | -1.48 (2.233) | -2.56 (2.352) | -2.45 (1.909) | -2.22 (2.887) | -2.14 (2.338)

4. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of OA to Week 12
Description: The PGA of OA was a 5-point Likert scale used to assess symptoms and activity impairment due to OA of the knee. Participants were asked to identify a number from 1 = "very good (asymptomatic and no limitation to normal activities)" to 5 = "very poor (very severe symptoms which are intolerable and inability to carry out all normal activities)" based on the question "Considering all the ways that OA of the knee affects you, how are you feeling today?". Change from baseline in PGA of OA to Week 12 is reported. A two-step multiple imputation procedure was used to address missing post-baseline scores.
Time Frame: Week 0 (Day 1; baseline) through Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 70
Unit on a scale | -0.34 (0.933) | -0.72 (1.123) | -0.81 (1.032) | -0.69 (1.377) | -0.57 (1.003)

5. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Over Time
Description: The WOMAC multiscale index is used to assess pain, stiffness, and joint functionality in the past 48 hours in participants with OA of the knee or hip. The WOMAC pain subscale consists of 5 questions assessing the participant's pain due to OA in the target knee. Each question was scored on an NRS scale from 0 to 10, and the WOMAC pain subscale score is calculated as the mean score from all 5 questions, where higher scores represent higher pain. Change from baseline in WOMAC pain subscale to Weeks 2, 4,6, 8, 10, and 18 is reported.
Time Frame: Baseline (Week 0; Day 1), Weeks 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), and 18 (Day 126)
Population: FAS included all randomized participants analyzed according to the intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 63 | 63 | 63 | 65 | 61
Unit on a scale
  Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  Week 2 | -1.32 (1.501) | -1.79 (1.988) | -1.58 (1.571) | -1.88 (1.953) | -1.30 (1.968)
  Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  Week 4 | -1.62 (1.635) | -2.33 (2.230) | -2.41 (1.939) | -2.60 (2.077) | -2.08 (2.000)
  Week 6: number analyzed (Participants) | 59 | 61 | 57 | 56 | 55
  Week 6 | -2.01 (1.541) | -2.76 (2.223) | -2.73 (1.852) | -3.07 (2.065) | -2.40 (2.114)
  Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  Week 8 | -2.01 (1.840) | -2.96 (2.259) | -2.91 (1.954) | -3.33 (1.964) | -2.56 (2.431)
  Week 10: number analyzed (Participants) | 53 | 56 | 52 | 48 | 46
  Week 10 | -2.14 (1.886) | -3.22 (2.282) | -2.89 (2.052) | -3.54 (2.055) | -2.89 (2.283)
  Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  Week 18 | -2.00 (2.090) | -3.02 (2.388) | -2.61 (2.107) | -3.50 (1.988) | -2.97 (2.219)

6. Secondary Outcome: Change From Baseline in WOMAC PF Subscale Over Time
Description: The WOMAC multiscale index is used to assess pain, stiffness, and joint functionality in the past 48 hours in participants with OA of the knee or hip. The WOMAC PF subscale consists of 17 questions assessing the participant's difficulty in performing activities of daily living due to OA in the target knee. Each question is scored on an NRS scale from 0 to 10, and the WOMAC PF subscale score is calculated as the mean score from all 17 questions, where higher scores represent worse function. Change from baseline in WOMAC physical function to Weeks 2, 4, 6, 8, 10, and 18 is reported.
Time Frame: Baseline (Week 0; Day 1), Weeks 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), and 18 (Day 126)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 63 | 63 | 63 | 65 | 61
Unit on a scale
  Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  Week 2 | -1.06 (1.621) | -1.64 (1.877) | -1.56 (1.417) | -1.80 (1.778) | -0.96 (1.728)
  Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  Week 4 | -1.59 (1.812) | -2.07 (1.933) | -2.20 (1.701) | -2.39 (2.062) | -1.62 (1.708)
  Week 6: number analyzed (Participants) | 59 | 61 | 57 | 56 | 55
  Week 6 | -1.77 (1.670) | -2.43 (1.946) | -2.43 (1.436) | -2.71 (2.001) | -1.92 (1.945)
  Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  Week 8 | -1.64 (1.856) | -2.82 (1.960) | -2.68 (1.792) | -3.06 (1.858) | -2.06 (2.114)
  Week 10: number analyzed (Participants) | 53 | 56 | 52 | 48 | 46
  Week 10 | -1.74 (1.994) | -2.85 (1.944) | -2.65 (1.671) | -3.30 (1.979) | -2.26 (2.063)
  Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  Week 18 | -1.55 (2.267) | -2.71 (2.141) | -2.37 (1.722) | -3.17 (1.812) | -2.24 (1.810)

7. Secondary Outcome: Change From Baseline in WOMAC Overall Score Over Time
Description: The WOMAC overall score consisted of all 24 questions reported in the WOMAC questionnaire to assess: i) pain subscale, ii) PF subscale and iii) stiffness subscale. WOMAC overall score was calculated as the mean score from all 24 questions each scored on a Likert scale from 0 to 10 where higher scores represent worse outcome. Change from baseline in weekly average of WOMAC overall score to Weeks 2, 4, 6, 8, 10, 12, and 18 is reported.
Time Frame: Baseline (Week 0; Day 1), Weeks 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 64 | 63 | 64 | 65 | 61
Unit on a scale
  Week 2: number analyzed (Participants) | 64 | 63 | 64 | 65 | 58
  Week 2 | -1.11 (1.546) | -1.71 (1.836) | -1.58 (1.343) | -1.88 (1.735) | -1.04 (1.695)
  Week 4: number analyzed (Participants) | 58 | 61 | 60 | 59 | 61
  Week 4 | -1.66 (1.706) | -2.14 (1.958) | -2.25 (1.667) | -2.45 (2.000) | -1.74 (1.671)
  Week 6: number analyzed (Participants) | 59 | 62 | 57 | 57 | 56
  Week 6 | -1.85 (1.583) | -2.54 (1.968) | -2.52 (1.426) | -2.79 (1.951) | -1.98 (1.984)
  Week 8: number analyzed (Participants) | 54 | 56 | 58 | 49 | 46
  Week 8 | -1.75 (1.792) | -2.85 (1.995) | -2.69 (1.757) | -3.12 (1.822) | -2.19 (2.102)
  Week 10: number analyzed (Participants) | 53 | 56 | 52 | 48 | 46
  Week 10 | -1.86 (1.907) | -2.94 (1.995) | -2.72 (1.663) | -3.35 (1.954) | -2.43 (2.022)
  Week 12: number analyzed (Participants) | 47 | 54 | 52 | 41 | 42
  Week 12 | -1.82 (1.945) | -3.00 (2.087) | -2.76 (1.616) | -3.48 (2.121) | -2.56 (1.956)
  Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  Week 18 | -1.68 (2.148) | -2.78 (2.153) | -2.46 (1.718) | -3.24 (1.784) | -2.42 (1.767)

8. Secondary Outcome: Change From Baseline in WOMAC Stiffness Scores Over Time
Description: The WOMAC stiffness function subscale consists of 2 questions assessing stiffness due to OA in the target knee. Stiffness is defined as a sensation of decreased ease of movement in the target knee. Each question is scored on an NRS scale from 0 to 10, and the WOMAC stiffness function subscale score is calculated as the mean score from the 2 questions, where higher scores represent higher stiffness. Change from baseline in WOMAC stiffness score to Weeks 2, 4, 6, 8, 10, 12, and 18 is reported.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 64 | 63 | 64 | 65 | 61
Unit on a scale
  Week 2: number analyzed (Participants) | 64 | 63 | 64 | 65 | 58
  Week 2 | -1.30 (1.887) | -2.06 (2.015) | -1.85 (1.927) | -2.13 (2.020) | -0.99 (1.805)
  Week 4: number analyzed (Participants) | 58 | 61 | 60 | 59 | 61
  Week 4 | -1.88 (1.938) | -2.26 (2.146) | -2.33 (2.127) | -2.55 (2.368) | -1.91 (2.009)
  Week 6: number analyzed (Participants) | 59 | 62 | 57 | 57 | 56
  Week 6 | -2.13 (1.837) | -2.79 (2.307) | -2.72 (1.871) | -2.97 (2.428) | -2.27 (2.314)
  Week 8: number analyzed (Participants) | 54 | 56 | 58 | 49 | 46
  Week 8 | -1.99 (2.125) | -2.85 (2.260) | -2.85 (2.103) | -3.07 (2.104) | -2.39 (2.633)
  Week 10: number analyzed (Participants) | 53 | 56 | 52 | 48 | 46
  Week 10 | -2.13 (2.060) | -2.99 (2.277) | -2.96 (1.977) | -3.29 (2.091) | -2.67 (2.329)
  Week 12: number analyzed (Participants) | 47 | 54 | 52 | 41 | 42
  Week 12 | -2.29 (2.034) | -3.06 (2.380) | -3.06 (2.040) | -3.43 (2.407) | -2.85 (2.372)
  Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  Week 18 | -2.04 (2.192) | -2.76 (2.401) | -2.86 (1.988) | -3.17 (1.797) | -2.62 (2.152)

9. Secondary Outcome: Change From Baseline in PGA of OA Over Time
Description: The PGA of OA was a 5-point Likert scale used to assess symptoms and activity impairment due to OA of the knee. Participants were asked to identify a number from 1 = "very good (asymptomatic and no limitation to normal activities)" to 5 = "very poor (very severe symptoms which are intolerable and inability to carry out all normal activities)" based on the question "Considering all the ways that OA of the knee affects you, how are you feeling today?". Change from baseline in PGA of OA to Weeks 2, 4, 8, 10, and 18 is reported.
Time Frame: Baseline, Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 10 (Day 70), and 18 (Day 126)
Population: FAS included all randomized participants analyzed according to the intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure. Number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 62 | 62 | 60 | 65 | 60
Unit on a scale
  Week 2: number analyzed (Participants) | 62 | 62 | 60 | 65 | 57
  Week 2 | -0.35 (0.812) | -0.56 (0.917) | -0.67 (0.933) | -0.42 (1.059) | -0.37 (0.698)
  Week 4: number analyzed (Participants) | 56 | 60 | 57 | 59 | 60
  Week 4 | -0.48 (0.738) | -0.68 (1.066) | -0.86 (1.043) | -0.86 (1.106) | -0.48 (0.792)
  Week 8: number analyzed (Participants) | 53 | 55 | 54 | 49 | 45
  Week 8 | -0.57 (0.910) | -0.80 (1.026) | -1.02 (1.090) | -1.04 (1.098) | -0.51 (0.843)
  Week 10: number analyzed (Participants) | 52 | 55 | 49 | 48 | 45
  Week 10 | -0.42 (0.723) | -0.76 (0.922) | -1.02 (1.010) | -1.06 (1.295) | -0.67 (0.826)
  Week 18: number analyzed (Participants) | 44 | 50 | 48 | 39 | 43
  Week 18 | -0.39 (0.655) | -0.66 (1.022) | -0.83 (1.117) | -1.10 (1.294) | -0.56 (0.700)

10. Secondary Outcome: Percentage of Responder Participants Measured by Osteoarthritis Research Society International (OARSI) Responder Index Using Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Definition
Description: The OMERACT-OARSI responder index is calculated from the WOMAC Pain subscale, the WOMAC Physical Function Subscale and the PGA of OA. A participant is classified as a responder if: 1. >= 2-point absolute change from Baseline to Week X or a >= 50% improvement is reported in the WOMAC Pain or the PF subscales; 2. At least 2 of the following 3 conditions are true: >= 1-point absolute change from Baseline to Week X or >= 20% improvement is reported in the WOMAC Pain subscale, >= 1-point absolute change from Baseline to Week X or >= 20% improvement is reported in the WOMAC PF subscale or >= 1-point absolute change from Baseline to Week X is reported in the PGA of OA. Percentage of responder participants are reported.
Time Frame: Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 65 | 64 | 68 | 67 | 65
Percentage of participants
  Week 2: number analyzed (Participants) | 65 | 64 | 68 | 67 | 64
  Week 2 | 47.7 | 62.5 | 61.8 | 59.7 | 40.6
  Week 4: number analyzed (Participants) | 59 | 62 | 64 | 61 | 65
  Week 4 | 59.3 | 67.7 | 73.4 | 65.6 | 63.1
  Week 8: number analyzed (Participants) | 56 | 57 | 60 | 51 | 51
  Week 8 | 58.9 | 80.7 | 80.0 | 86.3 | 68.6
  Week 12: number analyzed (Participants) | 49 | 55 | 55 | 42 | 46
  Week 12 | 59.2 | 80.0 | 80.0 | 85.7 | 67.4
  Week 18: number analyzed (Participants) | 47 | 52 | 54 | 41 | 47
  Week 18 | 55.3 | 78.8 | 72.2 | 80.5 | 70.2

11. Secondary Outcome: Percentage of Participants With Improvement of >= 2 Points in PGA of OA
Description: The PGA of OA was a 5-point Likert scale used to assess symptoms and activity impairment due to OA of the knee. Participants were asked to identify a number from 1 = "very good (asymptomatic and no limitation to normal activities)" to 5 = "very poor (very severe symptoms which are intolerable and inability to carry out all normal activities)" based on the question "Considering all the ways that OA of the knee affects you, how are you feeling today?". Percentage of participants with improvement of >= 2 points in PGA of OA at Weeks 2, 4, 8, 12, and 18 is reported.
Time Frame: Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 62 | 62 | 60 | 65 | 60
Percentage of participants
  Week 2: number analyzed (Participants) | 62 | 62 | 60 | 65 | 57
  Week 2 | 9.7 | 9.7 | 16.7 | 12.3 | 7.0
  Week 4: number analyzed (Participants) | 56 | 60 | 57 | 59 | 60
  Week 4 | 8.9 | 26.7 | 24.6 | 22.0 | 6.7
  Week 8: number analyzed (Participants) | 53 | 55 | 54 | 49 | 45
  Week 8 | 17.0 | 23.6 | 25.9 | 28.6 | 4.4
  Week 12: number analyzed (Participants) | 46 | 53 | 49 | 40 | 41
  Week 12 | 10.9 | 18.9 | 20.4 | 32.5 | 7.3
  Week 18: number analyzed (Participants) | 44 | 50 | 48 | 39 | 43
  Week 18 | 2.3 | 20.0 | 22.9 | 25.6 | 4.7

12. Secondary Outcome: Change From Baseline in Weekly Average of Daily NRS Pain Score Over Time
Description: The NRS is an 11-point Likert scale used to assess pain, where participants were asked to describe their average pain in the target knee by identifying a number from 0 = "no pain" to 10 = "most severe pain imaginable over the previous 24 hours". This will be recorded on a daily basis at approximately the same time every morning via ePRO diary. Change from baseline in weekly average of daily NRS to Weeks 2, 4, 6, 8, 10, and 18 is reported.
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), and 18 (Day 126)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 66 | 64 | 65 | 66 | 65
Unit on a scale
  Week 2 | -1.62 (1.704) | -1.86 (1.949) | -1.97 (2.012) | -2.26 (2.129) | -1.10 (1.811)
  Week 4: number analyzed (Participants) | 61 | 64 | 64 | 65 | 64
  Week 4 | -1.88 (1.653) | -2.50 (2.163) | -2.68 (2.177) | -2.65 (2.333) | -1.66 (1.854)
  Week 6: number analyzed (Participants) | 62 | 63 | 61 | 57 | 58
  Week 6 | -2.17 (1.687) | -2.83 (2.248) | -3.00 (2.192) | -3.35 (2.498) | -1.97 (2.020)
  Week 8: number analyzed (Participants) | 55 | 59 | 61 | 52 | 52
  Week 8 | -2.27 (1.736) | -2.91 (2.084) | -3.09 (2.205) | -3.45 (2.365) | -2.18 (2.274)
  Week 10: number analyzed (Participants) | 55 | 55 | 56 | 51 | 46
  Week 10 | -2.38 (2.001) | -3.18 (1.930) | -3.24 (2.294) | -3.57 (2.274) | -2.28 (2.047)
  Week 18: number analyzed (Participants) | 42 | 48 | 52 | 38 | 44
  Week 18 | -2.08 (2.120) | -3.18 (2.237) | -2.90 (2.157) | -3.63 (2.383) | -2.45 (1.969)

13. Secondary Outcome: Percentage of Participants With >= 30% and >= 50% Reductions in Weekly Average of Daily NRS Pain Score Over Time
Description: The NRS is an 11-point Likert scale used to assess pain, where participants were asked to describe their average pain in the target knee by identifying a number from 0 = "no pain" to 10 = "most severe pain imaginable over the previous 24 hours". This will be recorded on a daily basis at approximately the same time every morning via ePRO diary. Percentage of participants with >= 30% and >= 50% reductions in weekly average of daily NRS pain score are reported.
Time Frame: Baseline (Day -7 to Day -1, inclusive), Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 66 | 64 | 65 | 66 | 65
Percentage of participants
  >=30%: Week 2 | 34.8 | 34.4 | 41.5 | 43.9 | 21.5
  >=30%: Week 4: number analyzed (Participants) | 61 | 64 | 64 | 65 | 64
  >=30%: Week 4 | 47.5 | 50.0 | 64.1 | 53.8 | 29.7
  >=30%: Week 8: number analyzed (Participants) | 55 | 59 | 61 | 52 | 52
  >=30%: Week 8 | 56.4 | 67.8 | 67.2 | 61.5 | 42.3
  >=30%: Week 12: number analyzed (Participants) | 50 | 55 | 55 | 44 | 46
  >=30%: Week 12 | 58.0 | 76.4 | 65.5 | 72.7 | 47.8
  >=30%: Week 18: number analyzed (Participants) | 42 | 48 | 52 | 38 | 44
  >=30%: Week 18 | 42.9 | 72.9 | 67.3 | 65.8 | 54.5
  >=50%: Week 2 | 15.2 | 25.0 | 29.2 | 30.3 | 13.8
  >=50%: Week 4: number analyzed (Participants) | 61 | 64 | 64 | 65 | 64
  >=50%: Week 4 | 24.6 | 32.8 | 40.6 | 36.9 | 15.6
  >=50%: Week 8: number analyzed (Participants) | 55 | 59 | 61 | 52 | 52
  >=50%: Week 8 | 32.7 | 45.8 | 54.1 | 57.7 | 26.9
  >=50%: Week 12: number analyzed (Participants) | 50 | 55 | 55 | 44 | 46
  >=50%: Week 12 | 44.0 | 54.5 | 49.1 | 54.5 | 26.1
  >=50%: Week 18: number analyzed (Participants) | 42 | 48 | 52 | 38 | 44
  >=50%: Week 18 | 26.2 | 54.2 | 50.0 | 52.6 | 29.5

14. Secondary Outcome: Percentage of Participants With >= 30% and >= 50% Reductions in WOMAC Pain Subscale Score Over Time
Description: The WOMAC multiscale index is used to assess pain, stiffness, and joint functionality in the past 48 hours in participants with OA of the knee or hip. The WOMAC pain subscale consists of 5 questions assessing the participant's pain due to OA in the target knee. Each question was scored on an NRS scale from 0 to 10, and the WOMAC pain subscale score is calculated as the mean score from all 5 questions, where higher scores represent higher pain. Percentage of participants with >= 30% and >= 50% reductions in WOMAC pain subscale score over time are reported.
Time Frame: Baseline (Week 0; Day 1), Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 63 | 63 | 63 | 65 | 61
Percentage of participants
  >=30%: Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  >=30%: Week 2 | 30.2 | 39.7 | 36.5 | 50.8 | 24.1
  >=30%: Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  >=30%: Week 4 | 40.4 | 54.1 | 61.7 | 61.0 | 47.5
  >=30%: Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  >=30%: Week 8 | 55.6 | 64.3 | 64.9 | 71.4 | 56.5
  >=30%: Week 12: number analyzed (Participants) | 47 | 54 | 52 | 40 | 42
  >=30%: Week 12 | 59.6 | 68.5 | 67.3 | 75.0 | 66.7
  >=30%: Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  >=30%: Week 18 | 51.1 | 70.6 | 62.7 | 76.9 | 69.8
  >=50%: Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  >=50%: Week 2 | 14.3 | 23.8 | 17.5 | 33.8 | 10.3
  >=50%: Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  >=50%: Week 4 | 24.6 | 31.1 | 40.0 | 55.9 | 26.2
  >=50%: Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  >=50%: Week 8 | 35.2 | 46.4 | 49.1 | 57.1 | 34.8
  >=50%: Week 12: number analyzed (Participants) | 47 | 54 | 52 | 40 | 42
  >=50%: Week 12 | 31.9 | 51.9 | 50.0 | 62.5 | 42.9
  >=50%: Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  >=50%: Week 18 | 33.3 | 51.0 | 43.1 | 59.0 | 41.9

15. Secondary Outcome: Percentage of Participants With >= 30% and >= 50% Reductions in WOMAC Physical Function Subscale Over Time
Description: The WOMAC PF subscale consists of 17 questions assessing the participant's difficulty in performing activities of daily living due to OA in the target knee. Each question is scored on an NRS scale from 0 to 10, and the WOMAC PF subscale score is calculated as the mean score from all 17 questions, where higher scores represent worse function. Percentage of participants with >= 30% and >= 50% reductions in WOMAC physical function subscale over time are reported.
Time Frame: Baseline (Week 0; Day 1), Weeks 2 (Day 14), 4 (Day 28), 8 (Day 56), 12 (Day 84), and 18 (Day 126)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 63 | 63 | 63 | 65 | 61
Percentage of participants
  >=30%: Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  >=30%: Week 2 | 30.2 | 42.9 | 39.7 | 47.7 | 22.4
  >=30%: Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  >=30%: Week 4 | 47.4 | 52.5 | 61.7 | 59.3 | 37.7
  >=30%: Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  >=30%: Week 8 | 50.0 | 64.3 | 63.2 | 69.4 | 47.8
  >=30%: Week 12: number analyzed (Participants) | 47 | 54 | 52 | 40 | 42
  >=30%: Week 12 | 42.6 | 72.2 | 67.3 | 72.5 | 54.8
  >=30%: Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  >=30%: Week 18 | 42.2 | 72.5 | 64.7 | 74.4 | 60.5
  >=50%: Week 2: number analyzed (Participants) | 63 | 63 | 63 | 65 | 58
  >=50%: Week 2 | 14.3 | 22.2 | 23.8 | 33.8 | 12.1
  >=50%: Week 4: number analyzed (Participants) | 57 | 61 | 60 | 59 | 61
  >=50%: Week 4 | 28.1 | 31.1 | 41.7 | 54.2 | 19.7
  >=50%: Week 8: number analyzed (Participants) | 54 | 56 | 57 | 49 | 46
  >=50%: Week 8 | 33.3 | 51.8 | 47.4 | 57.1 | 26.1
  >=50%: Week 12: number analyzed (Participants) | 47 | 54 | 52 | 40 | 42
  >=50%: Week 12 | 34.0 | 46.3 | 50.0 | 62.5 | 35.7
  >=50%: Week 18: number analyzed (Participants) | 45 | 51 | 51 | 39 | 43
  >=50%: Week 18 | 33.3 | 45.1 | 39.2 | 59.0 | 34.9

16. Secondary Outcome: Serum Concentration of MEDI7352
Description: Serum concentration of MEDI7352 is reported.
Time Frame: Baseline (Day 1), Day 7; pre-dose on Days 14, 28, 42, 56, and 70; and on Days 74, 77, 84, 126, and 224
Population: Pharmacokinetic (PK) analysis set included participants who received at least one dose of double-blind study treatment per the protocol for whom any post-baseline PK data are available and who did not violate or deviate from the protocol in ways that would significantly affect the PK analyses. Number of participants analyzed (N) denotes those participants who were analyzed for this outcome measure. Number analyzed (n) denotes those participants who had adequate serum samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4
Number analyzed (Participants) | 70 | 68 | 67 | 68
ng/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7: number analyzed (Participants) | 63 | 62 | 66 | 65
  Day 7 | 326.863 (98.989) | 681.322 (159.914) | 2149.062 (109.2763) | 3582.265 (364.200)
  Day 14: number analyzed (Participants) | 65 | 63 | 67 | 67
  Day 14 | 50.337 (538.604) | 144.242 (475.607) | 379.882 (488.933) | 650.864 (624.642)
  Day 28: number analyzed (Participants) | 57 | 58 | 62 | 56
  Day 28 | 11.025 (853.538) | 28.332 (2745.856) | 43.644 (6705.491) | 222.665 (3963.855)
  Day 42: number analyzed (Participants) | 55 | 54 | 59 | 50
  Day 42 | 5.895 (846.517) | 12.375 (2578.767) | 30.005 (11978.840) | 116.951 (14993.947)
  Day 56: number analyzed (Participants) | 0 | 53 | 58 | 51
  Day 56 |  | 6.625 (2133.678) | 20.546 (13626.951) | 85.779 (15987.305)
  Day 70: number analyzed (Participants) | 0 | 0 | 55 | 44
  Day 70 |  |  | 17.124 (15147.088) | 57.042 (18183.372)
  Day 74: number analyzed (Participants) | 48 | 53 | 55 | 42
  Day 74 | 10.943 (1833.135) | 22.074 (4305.129) | 116.544 (25316.322) | 551.099 (18558.506)
  Day 77: number analyzed (Participants) | 45 | 50 | 52 | 44
  Day 77 | 5.011 (1322.708) | 9.356 (3099.752) | 47.108 (39692.068) | 271.511 (36387.885)
  Day 84: number analyzed (Participants) | 0 | 0 | 56 | 45
  Day 84 |  |  | 10.482 (6086.596) | 43.062 (13640.856)
  Day 126: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 224: number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to MEDI7352
Description: Number of participants with ADA to MEDI7352 are reported. Treatment-induced ADA positive is defined as ADA negative at baseline and positive at least 1 post-baseline ADA assessment. Treatment-boosted ADA positive is defined as ADA positive at baseline, and the baseline titre is boosted by greater than the variability of the assay (commonly 4-fold) at >= 1 post-baseline timepoint. Persistent positive is defined as ADA negative at baseline and having at least 2 post-baseline ADA positive assessments (with >= 16 weeks between first and last positive) or ADA positive at last post-baseline assessment. Transiently positive is defined as ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: Baseline (Day 1), Day 7; pre-dose on Days 14, 28, 42, 56, and 70; and on Days 74, 77, 84, 126, and 224
Population: ADA evaluable participants included all participants in the safety analysis set who have a non-missing baseline and at least one non-missing post-baseline ADA results. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure. Number analyzed (n) denotes those participants who had adequate ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 66 | 67 | 67
Participants
  Treatment-induced ADA positive | 52 | 49 | 42 | 52 | 6
  Treatment-boosted ADA positive | 6 | 9 | 8 | 2 | 2
  Persistent positive ADA | 43 | 39 | 33 | 42 | 4
  Transiently positive ADA | 9 | 10 | 9 | 10 | 2

18. Secondary Outcome: ADA Titre in Participants Who Were ADA Positive at Baseline and/or Post-baseline
Description: The ADA titre in participants who were ADA positive at baseline and/or post-baseline is reported.
Time Frame: Baseline (Day 1), Day 7; pre-dose on Days 14, 28, 42, 56, and 70; and on Days 74, 77, 84, 126, and 224
Population: ADA evaluable participants included all participants in safety analysis set who have non-missing baseline and at least 1 non-missing post-baseline ADA results. Number of participants analyzed (N): number of participants who were ADA positive at baseline and/or post-baseline. Number analyzed (n): participants who had adequate ADA sample.
Measure: Median (Full Range); unit: Ratio
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 61 | 59 | 52 | 54 | 19
Ratio | 960.0 [30 to 122880] | 960.0 [30 to 245760] | 960.0 [30 to 15360] | 720.0 [30 to 122880] | 240.0 [30 to 3840]

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Population: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  Any TEAEs | 51 | 45 | 54 | 51 | 41
  Any TESAEs | 3 | 5 | 3 | 1 | 2

20. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination Reported as TEAEs
Description: Number of participants with clinically significant findings in physical examination reported as TEAE are reported. A physical examination included assessments of general appearance, skin, head and neck, examination of the oral cavity for any lesions, lymph nodes, thyroid, abdomen (bowel sounds, liver, and spleen palpation), back (including costovertebral angle tenderness), musculoskeletal/extremities, cardiovascular, and respiratory systems.
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants | 0 | 0 | 0 | 1 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings in Neurological Examination
Description: Number of participants with clinically significant abnormal findings in neurological examination is reported. The neurological examination included assessment of mental status, cranial nerves, motor examination (muscle strength and tone), upper and lower extremity deep tendon reflexes, plantar responses, sensory system examination, coordination, and gait.
Time Frame: Baseline (Day -45 to Day -1), Weeks 0 (Day 1), 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), 12 (Day 84), 18 (Day 126), 28 (Day 168), 32 (Day 224), and 36 (Day 252)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  Baseline | 0 | 0 | 0 | 0 | 0
  Week 0 | 0 | 0 | 0 | 0 | 0
  Week 2 | 1 | 0 | 0 | 0 | 0
  Week 4 | 0 | 0 | 0 | 0 | 1
  Week 6 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0
  Week 10 | 0 | 0 | 0 | 0 | 0
  Week 12 | 0 | 0 | 0 | 1 | 0
  Week 18 | 0 | 0 | 0 | 1 | 0
  Week 28 | 0 | 0 | 0 | 1 | 0
  Week 32 | 0 | 0 | 0 | 1 | 0
  Week 36 | 0 | 0 | 0 | 2 | 0

22. Secondary Outcome: Total Neuropathy Score-Nurse (TNSn) Over Time
Description: The TNSn, is a semiquantitative clinical assessment of peripheral nervous system function. The TNSn assessment is collected as scores of motor symptom, autonomic symptom, pin sensibility, sensory symptom, and vibration sensibility score. Each neuropathy item is scored on a 0 to 4 scale with total score ranging from 0 to 20. Higher total scores correlate with more severe neuropathy.
Time Frame: Baseline (Day -45 to Day -1), Weeks 0 (Day 1), 2 (Day 14), 4 (Day 28), 6 (Day 42), 8 (Day 56), 10 (Day 70), 12 (Day 84), 28 (Day 196), and 32 (Day 224)
Population: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 66 | 69 | 68 | 67
Unit on a scale
  Baseline: number analyzed (Participants) | 51 | 55 | 59 | 56 | 61
  Baseline | 1.5 (2.40) | 1.4 (1.94) | 1.0 (1.56) | 1.2 (1.69) | 1.5 (2.02)
  Week 0 | 1.3 (1.92) | 1.7 (2.26) | 1.4 (2.03) | 1.5 (2.29) | 1.8 (2.26)
  Week 2: number analyzed (Participants) | 66 | 65 | 69 | 67 | 65
  Week 2 | 1.1 (1.84) | 1.6 (2.42) | 1.2 (1.97) | 1.0 (1.70) | 1.5 (2.18)
  Week 4: number analyzed (Participants) | 61 | 64 | 64 | 64 | 65
  Week 4 | 1.0 (1.66) | 1.3 (1.98) | 0.9 (1.54) | 0.9 (1.61) | 1.4 (2.16)
  Week 6: number analyzed (Participants) | 61 | 62 | 62 | 60 | 61
  Week 6 | 1.0 (1.55) | 1.4 (2.23) | 0.9 (1.73) | 0.9 (1.48) | 1.5 (2.51)
  Week 8: number analyzed (Participants) | 56 | 57 | 62 | 52 | 52
  Week 8 | 1.0 (1.65) | 1.1 (1.86) | 0.6 (0.91) | 0.8 (1.62) | 1.2 (1.84)
  Week 10: number analyzed (Participants) | 56 | 56 | 55 | 51 | 50
  Week 10 | 1.1 (1.85) | 1.3 (2.06) | 0.8 (1.53) | 0.7 (1.20) | 1.1 (2.10)
  Week 12: number analyzed (Participants) | 48 | 58 | 59 | 52 | 49
  Week 12 | 0.9 (1.35) | 1.2 (1.88) | 0.8 (1.37) | 0.7 (1.23) | 1.1 (2.00)
  Week 28: number analyzed (Participants) | 6 | 9 | 8 | 10 | 9
  Week 28 | 1.7 (2.25) | 3.3 (2.69) | 2.5 (2.83) | 0.8 (0.92) | 2.9 (2.67)
  Week 32: number analyzed (Participants) | 41 | 49 | 51 | 43 | 48
  Week 32 | 1.5 (1.98) | 1.0 (1.50) | 0.5 (0.88) | 0.9 (1.64) | 1.0 (1.98)

23. Secondary Outcome: Change From Baseline in Weight (kg) to Week 12
Description: Change from baseline in weight (kg) to Week 12 is reported.
Time Frame: Baseline (Day -45 to -1) and Week 12
Population: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants evaluated at Week 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 66 | 66 | 65 | 66 | 64
kg | -0.25 (2.048) | 0.10 (2.343) | 0.34 (1.932) | -0.03 (1.864) | -0.34 (2.004)

24. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormalfinding in the vital sign parameters (body temperature, supine and standing blood pressure, pulse rate, and respiratory rate).
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  Bradycardia | 0 | 0 | 0 | 0 | 1
  Tachycardia | 1 | 0 | 0 | 0 | 0
  Tachycardia paroxysmal | 1 | 0 | 0 | 0 | 0
  Hypertension | 0 | 2 | 3 | 0 | 0
  Hypertensive crisis | 1 | 0 | 0 | 0 | 0
  Orthostatic hypotension | 1 | 1 | 1 | 0 | 1
  Pyrexia | 0 | 0 | 0 | 0 | 1

25. Secondary Outcome: Change From Baseline in Survey of Autonomic Symptoms (SAS) Total Impact Score
Description: The SAS is an instrument that measures autonomic symptoms used for assessing autonomic neuropathies in clinical trials. The SAS scale evaluates the presence of symptoms and the degree of severity. The SAS consists of 11 questions in women and 12 questions in men. Each question has a Yes or No answer to symptoms occurring 6 months prior to investigational product (IP) administration. Questions answered with "Yes" are further rated by asking the participant how much each symptom is bothering him or her. Each answer is scored on a scale from 1 to 5 where 1 = not at all and 5 = a lot, and a total symptom impact score is determined. The SAS total impact score is the total of the scores from each question (11 for women and 12 for men). The minimum score is 0 and the maximum is 55 for women and 60 for men. A higher score indicates worse autonomic dysfunction.
Time Frame: Baseline (Day 1; Week 0) and Day 252 (Week 36)
Population: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure. Number analyzed (n) denotes those participants who had adequate SAS impact score.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 40 | 42 | 44 | 38 | 44
Unit on a scale | -1.5 (4.78) | -1.1 (4.63) | -0.9 (4.13) | -1.6 (4.62) | -0.8 (3.50)

26. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs)
Description: Number of participants with clinically significant abnormal ECGs are reported.
Time Frame: Weeks 0 (Day 1), 2 (Day 14), 4 (Day 28), 8 (Day 56), 10 (Day 70), 12 (Day 84), 28 (Day 168), and 32 (Day 224)
Population: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure. Number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  Week 0 | 0 | 0 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 66 | 64 | 68 | 68 | 66
  Week 2 | 0 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 62 | 63 | 63 | 60 | 64
  Week 4 | 0 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 55 | 57 | 60 | 52 | 49
  Week 8 | 0 | 0 | 0 | 0 | 0
  Week 10: number analyzed (Participants) | 54 | 55 | 56 | 48 | 50
  Week 10 | 0 | 0 | 0 | 1 | 0
  Week 12: number analyzed (Participants) | 66 | 66 | 67 | 65 | 65
  Week 12 | 0 | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 8 | 10 | 11 | 10 | 9
  Week 28 | 0 | 0 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 48 | 50 | 54 | 45 | 49
  Week 32 | 0 | 0 | 1 | 0 | 1

27. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  COVID-19 | 16 | 5 | 10 | 12 | 8
  Anaemia | 0 | 1 | 1 | 0 | 0
  Leukopenia | 1 | 0 | 0 | 0 | 1
  Lymphopenia | 0 | 0 | 0 | 1 | 1
  Neutropenia | 0 | 0 | 0 | 1 | 1
  Hypercholesterolaemia | 1 | 0 | 1 | 1 | 0
  Hyperkalaemia | 0 | 2 | 0 | 0 | 0
  Hypertriglyceridaemia | 1 | 0 | 0 | 2 | 1
  Hypokalaemia | 0 | 0 | 1 | 0 | 1
  Hyponatraemia | 0 | 0 | 1 | 0 | 0
  Type 2 diabetes mellitus | 0 | 0 | 0 | 0 | 1
  Vitamin D deficiency | 0 | 1 | 0 | 0 | 0
  Glycosuria | 0 | 1 | 0 | 0 | 2
  Leukocyturia | 0 | 2 | 0 | 0 | 1
  Proteinuria | 0 | 0 | 2 | 0 | 2
  Activated partial thromboplastin time prolonged | 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 1
  Blood creatine phosphokinase increased | 2 | 1 | 1 | 0 | 2
  Blood folate decreased | 1 | 0 | 0 | 0 | 0
  Blood glucose increased | 0 | 1 | 0 | 1 | 0
  Blood uric acid increased | 0 | 0 | 0 | 1 | 0
  C-reactive protein increased | 1 | 0 | 0 | 1 | 0
  Coagulation factor increased | 1 | 0 | 0 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0 | 1
  Glycosylated haemoglobin increased | 1 | 0 | 0 | 0 | 0

28. Secondary Outcome: Change From Baseline in C-reactive Protein Level to Week 12
Description: Change from baseline in C-reactive protein level to Week 12 is reported.
Time Frame: Baseline (Day -7 to -1, inclusive) and Week 12
Population: FAS included all randomized participants analyzed according to the intent-to-treat principle whereby randomized study treatment will be analyzed regardless of the study treatment actually received. Number of participants analyzed (N) denotes the number of participants evaluated at Week 12.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 50 | 55 | 54 | 43 | 45
mg/L | -2.55 (1.975) | -3.34 (2.004) | -3.30 (2.422) | -3.68 (2.313) | -2.38 (1.971)

29. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Number of participants with injection site reactions are reported.
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants | 2 | 3 | 0 | 4 | 0

30. Secondary Outcome: Number of Participants With Abnormal X-ray and/or Magnetic Resonance Imaging (MRI) of Large Joints
Description: Number of participants with abnormal X-ray and/or MRI of large joints is reported.
Time Frame: Baseline (Day -45 to -1) and Week 32
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | MEDl7352 Dose Level 1 | MEDl7352 Dose Level 2 | MEDl7352 Dose Level 3 | MEDl7352 Dose Level 4 | Placebo
Number analyzed (Participants) | 70 | 68 | 69 | 68 | 69
Participants
  X-ray | 1 | 0 | 0 | 1 | 2
  MRI | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through 41 weeks (maximum observed duration)
Description: Safety analysis set included all participants who received at least 1 dose of any double-blind study drug and were analyzed according to the treatment they actually received.
Groups:
- MEDI7352 Dose Level 1: Participants received 6 doses of subcutaneous (SC) MEDl7352 Dose Level 1 injection once every 2 weeks (Q2W) during a 12-week parallel-group treatment period.
- MEDI7352 Dose Level 2: Participants received 6 doses of SC MEDl7352 Dose Level 2 injection Q2W during a 12-week parallel-group treatment period.
- MEDI7352 Dose Level 3: Participants received 6 doses of SC MEDl7352 Dose Level 3 injection Q2W during a 12-week parallel-group treatment period.
- MEDI7352 Dose Level 4: Participants received 6 doses of SC MEDl7352 Dose Level 4 injection Q2W during a 12-week parallel-group treatment period.
Arm/Group | MEDI7352 Dose Level 1 | MEDI7352 Dose Level 2 | MEDI7352 Dose Level 3 | MEDI7352 Dose Level 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/68 | 0/69 | 0/68 | 0/69
Serious Adverse Events (participants affected / at risk) | 3/70 | 5/68 | 3/69 | 1/68 | 2/69
Other Adverse Events (participants affected / at risk) | 51/70 | 45/68 | 54/69 | 51/68 | 40/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI7352 Dose Level 1 (N=70) | MEDI7352 Dose Level 2 (N=68) | MEDI7352 Dose Level 3 (N=69) | MEDI7352 Dose Level 4 (N=68) | Placebo (N=69)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of bladder sensation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI7352 Dose Level 1 (N=70) | MEDI7352 Dose Level 2 (N=68) | MEDI7352 Dose Level 3 (N=69) | MEDI7352 Dose Level 4 (N=68) | Placebo (N=69)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (7) | 4 (4) | 6 (7) | 5 (5) | 9 (11)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (6) | 2 (4) | 4 (6) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood folate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Accessory spleen (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulation factor increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug screen positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal calprotectin abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7) | 5 (5) | 3 (6) | 4 (4)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (3) | 5 (5) | 7 (9) | 3 (3)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Areflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 7 (8) | 9 (9) | 9 (11) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (4) | 0 (0)
Migraine (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (5) | 3 (4) | 2 (3) | 4 (5) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Resting tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial vein prominence (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Injection site erythema (General disorders) | 2 (2) | 6 (8) | 6 (7) | 9 (10) | 2 (2)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 5 (7) | 4 (5) | 1 (1) | 2 (2)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 2 (3) | 3 (4) | 0 (0) | 4 (7) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type iv hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 16 (16) | 5 (5) | 10 (10) | 12 (12) | 8 (8)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Concomitant medication and therapies data do not necessarily evaluate the safety and are therefore not considered as outcome measures in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04675034/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04675034/SAP_001.pdf